CLINICAL TRIAL: NCT06313411
Title: How do I Perform a Laparoscopic Removal of a Pelvic Retroperitoneal Schwannoma
Acronym: PRS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8778
Record Dates: First submitted 2023-12-14; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis Pelvic
Keywords: Endometriosis Pelvic; Schwannomas
MeSH Terms: conditions — Neurilemmoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Schwannomas are mainly benign tumors, which develop mainly in the skull or in the cervical region. Retroperitoneal location is rare, since it represents between 0.5 and 5% of scwhanomas. The malignant retroperitoneal form is, however, more common than in other locations.

Retroperitoneal schwannoma is often discovered during the exploration of unexplained lumbo-pelvic pain, or in the face of compression of nearby organs. Abdominopelvic CT and magnetic resonance imaging are essential to characterize the mass and verify its extension. The precise diagnosis is based on the pathological examination of the part, and complete surgical excision is the standard treatment.

Acquiring the surgical techniques and skills necessary to carry out these types of procedures is essential to providing optimal patient care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* suffering from symptomatic deep pelvic endometriosis
* having received treatment at the Strasbourg University Hospital during 2021 for a retro-peritoneal pelvic carcinoma
* having not expressed, after information, the reuse of their data for the purposes of this research.

Exclusion Criteria:

* Patient who expressed her opposition to participating in the study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: - Adult patient (≥18 years old) having received treatment at the Strasbourg University Hospital during 2021 for a retro-peritoneal pelvic carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
laparoscopic removal of a retroperitoneal pelvic schwannoma | Through study completion, an average of 1 month
  The aim of this research is to train surgeons to perform laparoscopic removal of a retroperitoneal pelvic schwanoma

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie Obstétrique - CHU de Strasbourg - France, Strasbourg, France